CLINICAL TRIAL: NCT02266459
Title: A Prospective, Open, Multicenter Study to Evaluate the Performance, Safety and Usability of the Microwave Technology Developed by Medfield Diagnostics When Collecting Measurement Data From Patients With Clinical Signs of Stroke.
Brief Title: Study to Evaluate Performance, Usability, Safety of Microwave Technology When Collecting Data From Patients With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medfield Diagnostics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MF04
Record Dates: First submitted 2014-10-13; First posted 2014-10-17 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Stroke; Healthy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Microwave technology (Medfield Diagnostics) — A microwave measurement will be performed. The procedure will take approximately 15 minutes (the duration of the actual measurements is < 1 minute) and will not interfere with the patient's standard of care at the Stroke Unit.

SUMMARY:
This is a prospective, open, multicenter study that will enroll patients admitted to and hospitalized at the Stroke Unit due to diagnosed stroke and healthy volunteers.

The main purpose of the study is to evaluate the ability of the Microwave Technology to deliver adequate measurement data.

DETAILED DESCRIPTION:
After written informed consent has been acquired a physical examination will be performed followed by confirmation of the inclusion/exclusion criteria. After subject enrollment the microwave measurement will be performed. The procedure will take approximately 15 minutes (the duration of the actual measurements is < 1 minute) and will not interfere with the patient's standard of care at the Stroke Unit.

The measurement data will be evaluated for the presence of signal artifacts. The diagnostic ability of the device will be evaluated using a leave-one-out cross validation method with the CT diagnosis as ground truth. Microwave signals are sensitive to the dielectric parameters of the investigated object. In biological matter this is often related to amount of water. Brain tissue has different dielectric properties from blood. The physiological changes inside the brain that occurs as a result of a stroke will change the dielectric parameters.

ELIGIBILITY:
Inclusion Criteria:

(Group A)

* Signed Informed Consent Form
* Patient diagnosed (by CT) with ischemic stroke, within 24 hours of stroke onset
* Patient should be ≥ 18 years of age

(Group B)

* Signed Informed Consent Form
* Patient diagnosed (by CT) with hemorrhagic stroke, within 48 hours of stroke onset
* Patient should be ≥ 18 years of age

(Group C)

* Signed Informed Consent Form
* Subject should be ≥ 18 years of age

Exclusion Criteria:

(Group A+B)

* Pregnant or nursing woman
* Woman of child bearing potential and not taking adequate contraceptive precautions
* Patient that has already received thrombolytic treatment
* Patient participating in any other clinical study that could interfere with the result in the present study
* Patient diagnosed with a condition associated with risk of poor protocol compliance
* Any other condition or symptoms preventing the patient from entering the study, according to the investigator´s judgment
* Any patient that according to the Declaration of Helsinki is deemed unsuitable for study enrollment

(Group C)

* Pregnant or nursing woman
* Woman of child bearing potential and not taking adequate contraceptive precautions
* Subject participating in any other clinical study that could interfere with the result in the present study
* Any other condition or symptoms preventing the subject from entering the study, according to the investigator´s judgment
* Any subject that according to the Declaration of Helsinki is deemed unsuitable for study enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2014-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Ability to deliver adequate measurement data | The procedure will take approximately 15 minutes
  To confirm that the device will deliver adequate measurement data for at least 80 % of the patients diagnosed with Hemorrhagic stroke and Ischemic stroke

SECONDARY OUTCOMES:
To confirm that the device will deliver adequate measurement data for at least 80 % of the healthy volunteers | The procedure will take approximately 15 minutes
Mean time (± standard deviation) needed to complete the measurement procedure for group A + B + C | The procedure will take approximately 15 minutes
To confirm the diagnostic ability of the device using a leave-one-out cross validation method | The procedure will take approximately 15 minutes
Occurrence of adverse events | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Erik Karlsson, MD, PhD, Principal Investigator — Sahlgrenska University hospital/Sahlgrenska, Dept. of Neurology
Locations (3):
- Sweden (3):
  - Strokeenheten, Södra Älvsborgs Sjukhus, Borås, Borås
  - Sahlgrenska University Hospital/Sahlgrenska, Dept. of Neurology, Gothenburg, Göteborg
  - Strokeenheten, Skaraborgs Sjukhus, Skövde